CLINICAL TRIAL: NCT04910295
Title: Immunogenicity and Safety of COVID-19 Vaccine in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Hun Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2013-121-1206
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Covid19
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: COVID-19 vaccine — Subjects will be vaccinated with COVID-19 vaccines approved in Korea. Data on specific vaccines will be gathered.

SUMMARY:
Serum antibody titre against COVID-19 spike protein will be measured before, after the first dose, and after the second dose (when applicable) in cancer patients who are receiving or received anti-cancer drugs. Side effects of vaccination and actual incidence of COVID-19 will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Patients who are receiving or received anti-cancer drugs
* Those who are not vaccinated against COVID-19 at the time of enrollment
* Written informed consent

Exclusion Criteria:

* Any contraindications to COVID-19 vaccines
* Those who were already vaccinated
* Those who are on immunosuppressants or infected with HIV
* Those who underwent organ transplantation
* Active infections (for example, pneumonia)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who are receiving or received anti-cancer drugs at Seoul National University Hospital, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Antibody titre after vaccination | 21-28 days after completion of vaccination
  Antibody titre as measured by Anti-SARS-CoV-2 ELISA (IgG)

SECONDARY OUTCOMES:
Antibody titer according to chemotherapy cycle, side effects, and use of corticosteroids or antipyretics | 21-28 days after completion of vaccination
  Antibody titre as measured by Anti-SARS-CoV-2 ELISA (IgG)
Incidence of COVID-19 infection | 6 months after completion of vaccination
  Incidence of actual COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing of IPD will be discussed and decided upon request.